CLINICAL TRIAL: NCT02285725
Title: Microdrilling Surgery for Full Thickness Chondral Lesions of the Knee Augmented With Concentrated Bone Marrow Aspirate, Platelet Rich Plasma and Hyaluronic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph E. Broyles (Other)
Responsible Party: Sponsor-Investigator, Joseph E. Broyles, Joseph E. Broyles, M.D., Bone and Joint Clinic of Baton Rouge
Organization: Bone and Joint Clinic of Baton Rouge (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMPRP1001
Record Dates: First submitted 2014-10-31; First posted 2014-11-07 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Unilateral Primary Osteoarthritis of Knee; Osteoarthritis Knee; Degeneration; Articular Cartilage, Knee; Degenerative Lesion of Articular Cartilage of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Augmented Microdrilling Surgery (Experimental)
  Interventions: Procedure: Microdrilling Surgery; Procedure: Injections of BMAC + PRP + HA

INTERVENTIONS:
Procedure: Microdrilling Surgery — All patients will undergo an arthroscopic surgical procedure in which small holes are drilled throughout the areas of damaged cartilage (standard of care)
Procedure: Injections of BMAC + PRP + HA — All patients will receive up to 12 intra-articular knee injections of BMAC (derived from iliac crest), PRP (derived from peripheral blood) and HA

SUMMARY:
This study seeks to evaluate a treatment for multiple full thickness chondral lesions in the knee. Eligible subjects will undergo a microdrilling surgery and up to 12 post operative intra-articular injections of bone marrow aspirate concentrate (BMAC), platelet rich plasma (PRP) and hyaluronic acid (HA).

ELIGIBILITY:
Inclusion Criteria: MRI-confirmed full-thickness unipolar or bipolar chondral lesion(s) from osteoarthritis.

Exclusion Criteria:

* Inflammatory arthritis
* Body mass index (BMI) greater than 35
* Presence of significant varus or valgus knee instability or unusually stiff knee
* Greater than 50% deviation of the mechanical axis
* Presence of active cardiac disease
* Presence of active pulmonary disease
* Prior septic arthritis of the involved joint
* Presence of active bacterial or Mycobacterial infection
* Presence of a known hypercoagulable state
* Pregnant or lactating females
* Subject known to be positive for hepatitis B, hepatitis C, or HIV
* Known allergy to hyaluronic acid
* Patients who are unable or unwilling to participate fully in post-operative physical therapy
* Patients with a contraindication to MRI scanning
* Any disorder that compromises ability to give consent or comply with study procedures
* Patients who are felt to be at significantly increased risk for elective orthopedic surgery
* Non-ambulatory patients
* Patients with cognitive impairment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change in International Knee Documentation Committee (IKDC) score | Change from baseline at 5 years post-operatively

SECONDARY OUTCOMES:
Joint Space Changes | 2 and 5 years post-operatively
  Evaluated by plain radiographs
MRI appearance of repair cartilage | 2 and 5 years post-operatively
  Evaluated using the MOCART scoring system
Frequency of adverse events requiring additional procedures | Continuously for 5 years post-operatively

REFERENCES:
- See also: Related Info — http://cartilageregenerationcenter.com